CLINICAL TRIAL: NCT00839553
Title: Intrapleural Minocycline After Manual Aspiration for the Prevention of Primary Spontaneous Pneumothorax. A Phase III Multicenter Prospective Randomized Controlled Trial
Brief Title: Intrapleural Minocycline After Aspiration of Spontaneous Pneumothorax
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: National Taiwan University Hospital (Other); Department of Health (Ambiguous)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 95042
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Pneumothorax
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Intrapleural Minocycline application

SUMMARY:
The estimated recurrence rate of primary spontaneous pneumothorax is 23-50% after the first episode, and the optimal treatment remains unknown. In the recently published British Thoracic Society (BTS) guidelines, simple aspiration is recommended as first line treatment for all primary pneumothoraces requiring intervention. However, the 1 year recurrence rate of this procedure was as high as 25-30%, making it inappropriate as a standard of care.

Intrapleural instillation of a chemical irritant (chemical pleurodesis) is an effective way to shorten the duration of air leaks and reduce the rates of recurrent spontaneous pneumothorax in surgical and non-surgical patients. Many chemical irritants (tetracycline, talc, and minocycline) have been used to decrease the rate of recurrence in spontaneous pneumothorax. Tetracycline, which was the most commonly used irritant, is no longer available. Talc insufflation of the pleural cavity is safe and effective for primary spontaneous pneumothorax. However, it should be applied either with surgical or medical thoracoscopy. Minocycline, a derivative of tetracycline, is as effective as tetracycline in inducing pleural fibrosis in rabbits. In the previous studies, we have shown that additional minocycline pleurodesis is a safe and convenient procedure to decrease the rates of ipsilateral recurrence after thoracoscopic treatment of primary spontaneous pneumothorax. In the present study, additional minocycline pleurodesis will be randomly administered in patients with first episode of primary spontaneous pneumothorax after simple aspiration. The primary goal is to test if intrapleural minocycline can reduce the rate of recurrence. The secondary goals are to evaluate the safety profile, short-term results, and long-term effects of minocycline pleurodesis after simple aspiration. The sites of study include National Taiwan University Hospital and Far Eastern Memorial Hospital. A total of 300 patients (150 patients in each arm) will be included for this study.

ELIGIBILITY:
Inclusion Criteria:

1. 15-50years old
2. primary pneumothorax first attack
3. viceral pleura to chest wall more then 2 cm on CXR

Exclusion Criteria:

1. the lungs unable to expad fully after aspiration
2. continuous leakage of air through chest tubes
3. status complicated with hemothorax
4. status post previous chest surgery or pleurodesis
5. patient unwilling to accept the trial

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-04; Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate

CONTACTS AND LOCATIONS:
Overall Officials: YC Lee, PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- Far Eastern Memorial Hospital, Banqiao District, Taipei, Taiwan